CLINICAL TRIAL: NCT01517334
Title: Multi-Center Phase 3 Trial of Minocycline HCl 1 mg Microspheres for the Use in Subjects With Peri-Implantitis: Clinical and Microbiological Evaluations
Brief Title: Arestin - Use in Subjects With Peri-Implantitis (With Subgingival Microbiological Evaluation)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OraPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-P-5266-M
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2014-04

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Treatment (minocycline HCl microspheres, 1mg) administered at Baseline (following randomization) and Day 90 to qualifying implant sites, plus full-mouth mechanical debridement (deep cleaning) at Baseline and Day 180.
  Interventions: Drug: Minocycline HCl Microspheres
- Control (No Intervention): Full-mouth mechanical debridement (deep cleaning) at Baseline and Day 180; no treatment

INTERVENTIONS:
Drug: Minocycline HCl Microspheres
  Other Names: Arestin (brand name)
  Arms: Treatment

SUMMARY:
The objective of the study is to evaluate the safety, effectiveness and anti-microbial effects of Arestin (minocycline HCl) 1 mg Microspheres in the treatment of subjects with peri-implantitis, when used in combination with mechanical debridement.

The hypothesis of the study is that Arestin in combination with mechanical debridement is more effective in the treatment of peri-implantitis when compared to mechanical debridement alone. The primary efficacy measure will be the reduction of probing depth at Day 180 as measured at qualifying implant sites.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of one osseointegrated implant with a diagnosis of peri-implantitis
* Absence of any significant oral soft tissue pathology
* At least one peri-implant site with an average of 2 probing depth readings between 5mm and 7mm (inclusive) when using a light force and with bleeding on probing within 30 seconds of the probing
* Confirmed evidence of pathologic bone loss
* At least 1mm of keratinized gingiva present around the implant

Exclusion Criteria:

* Pregnancy
* Allergy to tetracycline-class drug(s)
* Systemic medical condition(s) requiring antibiotic prophylaxis prior to invasive dental procedures
* Presence of active systemic infectious disease such as hepatitis, HIV, history of tuberculosis
* Diagnosis of clinically significant or unstable organic disease, or compromised healing potential
* Signs of untreated advanced periodontal disease and/or poor oral hygiene
* Subjects having a probing depth greater than 8mm at time of enrollment
* Subjects presenting with mobility of any dental implant
* Subjects having a qualifying implant under occlusal trauma or overloaded (as determined by the investigator)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in mean Probing Depth of qualifying implant sites | Baseline to Day 180

SECONDARY OUTCOMES:
Change in percentage of qualifying implants with Bleeding On Probing | Baseline to Day 180
Change in mean Probing Depth of qualifying implant sites | Baseline to Day 90
Change in percentage of qualifying implants with Bleeding on Probing | Baseline to Day 90

OTHER OUTCOMES:
Exploratory: Changes in proportions and numbers of red-complex bacteria (RCB) | Baseline to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS, Principal Investigator — University of North Carolina - Chapel Hill Dental School
Locations (10):
- United States (10):
  - University of Maryland, School of Dentistry, Baltimore, Maryland
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - University of Michigan - Michigan Center for Oral Health Research, Ann Arbor, Michigan
  - University of Missouri - Kansas City School of Dentistry Clinical Research Center, Kansas City, Missouri
  - University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina
  - University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina College of Dental Medicine, Charleston, South Carolina
  - UTHSC - College of Dentistry, Memphis, Tennessee
  - Virginia Commonwealth University School of Dentistry, Richmond, Virginia
  - Marquette University School of Dentstry, Milwaukee, Wisconsin